CLINICAL TRIAL: NCT00679458
Title: A Randomized, Double-blind, Cross-over Trial Comparing the Analgesic Potency and Side Effects of Buprenorphine and Ultra-low-dose Naloxone to Buprenorphine Alone
Brief Title: Randomized, Double-Blind Cross-Over Trial Of Buprenorphine and Low-Dose Naloxone Versus Buprenorphine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Indivior Inc. (Industry)
Responsible Party: Walter Ling, M.D., UCLA Integrated Substance Abuse Programs
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-06-005
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-11

CONDITIONS: Pain
Keywords: analgesia; pain; buprenorphine; opioid; naloxone
MeSH Terms: conditions — Pain; Agnosia | interventions — Buprenorphine; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. (Experimental): Study drug: buprenorphine and ultra-low-dose naloxone
  Interventions: Drug: buprenorphine and low-dose naloxone
- 2. (Active Comparator): Study drug: buprenorphine
  Interventions: Drug: buprenorphine alone

INTERVENTIONS:
Drug: buprenorphine and low-dose naloxone — each participant will be randomly assigned to order of study drug administration in a double-blind manner. Five doses of first study drug will be administered for 5 days, with each administration following the previous dose by not more than 2 days. Administration of the second study drug, buprenorphine only, will follow at least 2 days after the completion of the first study drug with the same administration criteria. Medication will be administered IV, and assessments will continue for 6 hours after administration. Study drugs include 1) buprenorphine 0.3mg and naloxone 0.02mg and, 2) buprenorphine 0.3mg.
  Arms: 1.
Drug: buprenorphine alone — each participant will be randomly assigned to order of study drug administration in a double-blind manner. Five doses of first study drug will be administered for 5 days, with each administration following the previous dose by not more than 2 days. Administration of the second study drug will follow at least 2 days after the completion of the first study drug with the same administration criteria. Medication will be administered IV, and assessments will continue for 6 hours after administration. Study drugs include 1) buprenorphine 0.3mg and naloxone 0.02mg and, 2) buprenorphine 0.3mg.
  Arms: 2.

SUMMARY:
This study compares two medications for analgesic potency and side effects in a sample of individuals with moderate pain. After screening, eligible participants will be randomly assigned to begin blinded treatment with one of two medications. Participants receive 5 daily doses of medication (no more than 2 days between each dose) followed by crossover to the opposite treatment condition for 5 additional daily doses. Each study day, participants will provide a daily pain assessment, receive administration of study medication, and will then be monitored and assessed for pain and side effects over 6 hours.

DETAILED DESCRIPTION:
Treatment of chronic pain typically relies on the effectiveness of opioid analgesics, however, side effects and the potential for users to develop tolerance and addiction may make physicians hesitant to prescribe them. The development of opioid analgesics with fewer side effects and decreased potential tolerance and addiction would increase the ability to safely and effectively treat pain. This study will determine whether the addition of an ultra-low dose of naloxone, an opioid antagonist, to buprenorphine, an opioid analgesic pain medication, increases the analgesic potency and reduces side effects compared to buprenorphine alone. Low doses of naloxone added to buprenorphine have been shown to increase the potency and reduce the side effects of buprenorphine in animal studies and in a human study with healthy volunteers. The current study aims to extend these findings by assessing the analgesic potency and side effects of a 15:1 ratio of buprenorphine to naloxone in a sample of 12 outpatient participants with moderate pain (4 or greater pain intensity) who are experienced with opioid analgesics. Participants will be randomly assigned to begin blinded treatment starting with one of two medication regimens: IV buprenorphine + ultra-low-dose naloxone or IV buprenorphine alone. Participants receive 5 daily doses of medication (no more than 2 days between each dose) followed by crossover to the opposite treatment condition for 5 additional daily doses. Each study day, participants will provide a daily pain assessment, receive administration of study medication, and will then be monitored and assessed for pain and side effects over the next six hours. Outcomes for the study include: (1) pain intensity as measured using the Brief Pain Inventory, pain intensity numerical rating scale, and the Beck Depression Inventory, and (2) self-reported side effects/adverse events. After completion of study participation, participants will resume pre-study pain treatments with their own physician.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following:

1. 18 years of age or older
2. Have chronic pain that is not related to cancer, defined as pain expected to last a month or more,(i.e. musculoskeletal pain or neuropathic pain)
3. Report pain of moderate to moderately-severe intensity during the week prior to the baseline screening visit (a score greater than or equal to 4 for average pain in the past week on the 0-10 point Pain Intensity-Numerical Rating Scale)
4. Have used prescription opioid and/or non-opioid analgesics for the pain on at least 15 of the 30 days prior to the initial baseline/screening visit and have clearance from their prescribing physician to discontinue all non-study-related opiates during study participation
5. Willing and able to comply with study procedures
6. Willing and able to provide written consent
7. If female, not pregnant or lactating and willing to use an acceptable method of birth control (e.g., condoms, IUD, birth control pills, or Depo-Provera)

Exclusion Criteria:

Participants must not meet any of the following:

1. Have a history of dependence on opiates, stimulants, alcohol, or benzodiazepines, as defined by DSM-IV criteria, within the past year (physical dependence on prescribed opioid analgesics is allowed but opioid dependence according to DSM-IV, i.e. opioid addiction, is not)
2. Use of any illicit or recreational drugs (heroin, cocaine, methamphetamine, marijuana, etc.) ; or use of any long-acting opioid (i.e., methadone) in the 30 days prior to the initial screening visit
3. Concomitant use of medications that are inhibitors of CYP3A4 (e.g., azole antifungals, macrolide antibiotics, and HIV protease inhibitors), or medications that induce CYP3A4 activity (e.g., anticonvulsants and rifampin) that may alter the metabolism of buprenorphine
4. Have a medical condition that, in the study physician's judgment, may interfere with safe study participation for the individual study candidate. Because medical conditions may differ in terms of safe participation on an individual basis, this criterion must be based on a physician's determination after a medical history, exam, and lab tests and may also involve consultation with a study candidate's primacy care physician. Some examples of medical conditions that may be exclusionary for a particular individual, however include active tuberculosis, unstable and/or significant cardiovascular or liver disease, unstable diabetes (i.e., glycosylated hemoglobin A1C of 12%), uncontrolled HIV infection, altered renal function (serum creatinine males and females:>3x upper limit of normal) or clinically significant elevated liver enzymes (ALT or AST greater than 3x the upper limit of normal)
5. Have a current neurological disorder (e.g., organic brain disease, dementia) or current major psychiatric disorder (e.g., schizophrenia, bipolar illness, or PTSD) that would make study agent compliance difficult, that would compromise informed consent, or that would jeopardize safety
6. Have a history of suicide attempts in the past 180 days and/or current serious suicidal risk
7. Have any history of a seizure disorder
8. Have a known allergy or sensitivity to buprenorphine or naloxone
9. Receiving long-acting opioids, such as methadone, LAAM, or sustained release morphine, for treatment of pain (due to problems with initiating buprenorphine treatment among patients receiving long-acting opioids)
10. Have recent surgery or a major medical procedure that could potentially interfere with study participation
11. Any other circumstances that, in the opinion of the investigators, would interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity | After each dose of study drug

SECONDARY OUTCOMES:
Self-reported side effects/adverse events | after each daily dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — UCLA Integrated Substance Abuse Programs
Locations (1):
- UCLA Integrated Substance Abuse Programs Outpatient Research Center, Los Angeles, California, United States